CLINICAL TRIAL: NCT00737919
Title: The Influence of Dietary Plant Sterols and Plant Stanols on Cholesterol and Plant Sterol Levels in Atheromatous Plaques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Professor Mauri Lepäntalo, Dept. of Surgery, Div of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215953
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2008-08

CONDITIONS: Atherosclerosis
Keywords: Cholesterol; Plant sterols; Atherosclerotic carotid plaques
MeSH Terms: conditions — Atherosclerosis | interventions — Sitosterols; Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): A group of subjects consuming daily 2 grams of plant stanols 4-6 weeks before the operation
  Interventions: Dietary Supplement: Plant Stanol
- 2 (Active Comparator): A group of patients consuming daily 2 grams of plant sterols 4-6 weeks before the operation
  Interventions: Dietary Supplement: Plant Sterol

INTERVENTIONS:
Dietary Supplement: Plant Stanol — Plant stanols in margarines daily 2 grams
  Arms: 1
Dietary Supplement: Plant Sterol — Plant sterols in margarines daily 2 grams
  Arms: 2

SUMMARY:
This study aims to explore whether the increased supply of dietary plant sterols and plant stanols have any influence on serum levels of phytosterols and on consistency of carotid atheromatous plaques.

DETAILED DESCRIPTION:
This is a double-blind randomized study. The study population will consist of 30 consecutive patients who will undergo an elective carotid endarterectomy due to a tight asymptomatic stenosis. The patients will be randomized into two groups consuming either plant sterol (2g/day) or plant stanol (2g/day) spreads for two to six weeks, until the operation. Serum lipids, lipoproteins and sterols will be analyzed at the randomization, before the operation and one month after the operation. The carotid arteries will be examined for their composition of sterols.

This study gives new information concerning the relationship between dietary consumption of plant sterols and stanols and the sterol composition of the carotid plaques.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic tight carotid plaques
* Age 40-80

Exclusion Criteria:

* No

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sterols in serum and carotid plaques at the operation | at operation and one month after operation

CONTACTS AND LOCATIONS:
Overall Officials: Tatu A. Miettinen, professor, Principal Investigator — Dept. of Medicine, Div. of Internal Medicine, Helsinki Univ. Central Hospital, Biomedicum Helsinki; Helena Gylling, Professor, Principal Investigator — Department of Clinical Nutrition, University of Kuopio and Kuopion University Central Hospital, Kuopio, Finland; Markku J Nissinen, MD, PhD, Principal Investigator — Dept. of Medicine, Div. of Gastroenterology, HUCH, Helsinki, Finland
Locations (1):
- Department of Surgery, Div. of Vascular Surgery, Helsinki University Central Hospital, Helsinki, Finland